CLINICAL TRIAL: NCT07219576
Title: PRISM: Phase 1b of Retifanlimab and Ruxolitinib In Solid Malignancies Progressing on Prior Checkpoint Inhibition
Brief Title: Retifanlimab and Ruxolitinib In Solid Malignancies
Acronym: PRISM
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Principal Investigator, Rana Mckay, Clinical Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 812209
Record Dates: First submitted 2025-10-20; First posted 2025-10-22 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Non Small Cell Lung Carcinoma; Renal Cell Carcinoma
Keywords: programmed death ligand-1 blocker; Janus kinase inhibitor; 3+3 dose escalation design; recommended phase 2 dose
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ruxolitinib plus retifanlimab (Experimental): Combination of the Janus kinase 1/2 inhibitor ruxolitinib plus the programmed cell death protein-1 blocker retifanlimab. The study utilizes a standard 3+3 dose escalation design evaluating 2 dose escalation levels (15 mg and 20 mg orally twice daily) and 2 dose de-escalation levels (10 mg and 5 mg orally twice daily, if necessary) of ruxolitinib with fixed dose retifanlimab (500 mg intravenously every 4 weeks), followed by an expansion cohort at the recommended phase 2 dose.
  Interventions: Drug: Ruxolitinib; Drug: Retifanlimab

INTERVENTIONS:
Drug: Ruxolitinib — Janus kinase 1/2 inhibitor
  Other Names: Jakafi; Jakavi
Drug: Retifanlimab — Programmed cell death protein-1 blocker
  Other Names: Zynyz

SUMMARY:
The goal of this clinical trial is to learn what dose of ruxolitinib can be given safely together with retifanlimab in patients with metastatic renal cell carcinoma and non-small cell lung carcinoma.

The main question it aims to answer is:

What is the maximum dose of ruxolitinib that can be used safely in patients with metastatic renal cell carcinoma and non-small cell lung carcinoma, and will it work?

Participants will:

Take drug ruxolitinib twice a day and keep a diary of when they take ruxolitinib at home; visit the clinic for infusions of retifanlimab every 4 weeks; visit the clinic for checkups and tests.

DETAILED DESCRIPTION:
The treatment landscape for renal cell carcinoma has evolved significantly with the use of immunotherapy. Immune checkpoint inhibitors are now used in both adjuvant and metastatic settings. Programmed cell death protein-1 (PD-1) inhibitors are utilized as adjuvant therapy following nephrectomy for high-risk disease, and in the metastatic setting as first-line treatment in combination with either cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) inhibition or vascular endothelial growth factor (VEGF) pathway blockade. Despite improvements in overall survival with these approaches, the majority of patients develop either intrinsic or acquired resistance, necessitating subsequent therapy. The optimal management of patients progressing on immunotherapy remains an important unmet need in renal cell carcinoma.

Also the therapeutic landscape for non-small cell lung cancer has been transformed by immunotherapy, with programmed cell death protein-1/programmed death-ligand 1 (PD-1/PD-L1) inhibitors now established as standard first-line therapy either as monotherapy for patients with high PD-L1 expression (≥50%) or in combination with chemotherapy regardless of PD-L1 status. Despite significant improvements in survival outcomes, most patients eventually develop resistance to PD-1/PD-L1 blockade. The optimal approach for non-small cell lung cancer progressing on immunotherapy remains unclear. The identification of effective treatment strategies for patients with immunotherapy-resistant non-small cell lung cancer represents a critical unmet need, particularly given the large patient population affected by this disease.

Ex vivo experiments by the investigators showed that Janus kinase inhibitors restore cytokine production and proliferation of exhausted T cells and that the Janus kinase 1/2 inhibitor ruxolitinib enhanced the efficacy of immune checkpoint inhibitors in cancer models. Also a preliminary clinical trial by the investigators showed encouraging results, inasmuch 10 of 19 evaluable patients responded to therapy with the Janus kinase 1/2 inhibitor ruxolitinib plus the programmed cell death protein-1 blocker nivolamab. Among the patients who responded, six had complete responses and additional two experienced an indeterminate response or stable disease.

Building on previous clinical trials, the investigators plan to use the Janus kinase 1/2 inhibitor ruxolitinib in combination with the PD-1 blocker retifanlimab in renal cell carcinoma and non-small cell lung cancer, two tumor types in which PD-1 blockers are effective at least in a subset of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced or metastatic clear cell renal cell carcinoma or non-small cell lung carcinoma having progressed on prior PD-1/PD-L1 therapy (radiographic progression within 6 months of discontinuing immunotherapy; immunotherapy does not need to be the immediate line of preceding therapy).
2. Decline standard of care treatment or no available standard of care treatment.
3. Measurable disease per Response Evaluation Criteria in Solid Tumors version 1.1.
4. Eastern Cooperative Oncology Group performance status of 0 or 1.
5. Adequate organ and marrow function:

   * Absolute neutrophil count ≥ 1.0×10^9/L.
   * Platelet count ≥ 100×10^9/L.
   * Hemoglobin level ≥ 8.5 g/dL; criteria must be met without erythropoietin dependency and without packed red blood cell transfusion within the last 2 weeks.
   * Serum creatinine ≤ 2 mg/dL (or estimated creatinine clearance ≥ 30 mL/minute calculated by the Cockcroft Gault or Modification of Diet in Renal Disease formulas).
   * Aspartate Aminotransferase and Alanine Aminotransferase ≤ 2.5 x upper limit of normal.
   * Bilirubin ≤1.5 x upper limit of normal.
6. Ability to take oral medication and be willing to adhere to the study intervention.
7. Willingness to comply with all study procedures and availability for the duration of the study.

Exclusion Criteria:

1. Pregnancy or lactation.
2. No prior treatment with Janus kinase inhibitors.
3. No more than one prior line of PD-1/PD-L1 therapy. No limit on prior lines of systemic therapy. PD-1/PD-L1 therapy does not need to be the most immediate prior line of therapy. Patients with progressive disease as best response to prior PD-1/PD-L1 therapy are not eligible. Need to have either stable disease, partial response, or complete response as best response using RECIST version 1.1 principles to prior PD-1/PD-L1 therapy.
4. Received systemic anti-cancer therapy within 3 weeks of enrollment or small molecule kinase inhibitors within two weeks or six elimination half-lives of enrollment, whichever is sooner.
5. Has received prior radiotherapy within one week before enrollment.
6. Has had history of major surgery less than two weeks before enrollment. Adequate wound healing after major surgery must be assessed clinically.
7. Failure to recover from any immune related adverse event from prior immunotherapy to Common Terminology Criteria in Adverse Event grade ≤ 1 (participants with grade ≤ 2 sensory neuropathy, endocrinopathies controlled by hormone replacement, or other grade ≤ 2 not constituting a safety risk based on investigator's judgment are eligible).
8. Known active central nervous system metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate, provided they are clinically stable and without the requirement of steroid treatment for at least 14 days prior to enrollment.
9. Known active or history of autoimmune disease that requires steroids or immunosuppressive agents. Patients are allowed in the study if they have vitiligo, type 1 diabetes mellitus, controlled asthma; residual hypo- or hyperthyroidism due to an autoimmune condition not requiring immunosuppressive treatment; psoriasis, atopic dermatitis, or another autoimmune skin condition that is managed without steroids or immunosuppressive agents; or arthritis that is managed without systemic therapy beyond oral acetaminophen and non-steroidal anti-inflammatory drugs.
10. Diagnosis of immunodeficiency or receiving systemic steroid therapy (equivalent of prednisone > 10 mg daily) or any other form of immunosuppressive therapy within seven days prior to the first dose of study treatment. The use of physiologic doses of corticosteroids is permitted. Intra-articular, intra-ocular, intra-nasal, inhalation and ocular steroids are permitted.
11. Active infections requiring systemic antibiotics or antifungal or antiviral treatment within 7 days before first dose of study treatment.
12. Active tuberculosis.
13. Active immunodeficiency virus (HIV) infection. To be enrolled, patients with history of HIV must have an undetectable viral load at screening.
14. Active hepatitis B or hepatitis C virus infections. To be enrolled, patients with a history of these infections must have been treated and cured with undetectable viral load at screening.
15. Have clinically significant cardiovascular disease defined as:

    * Cerebral vascular accident/stroke or myocardial infarction (<6 months prior to enrollment)
    * Unstable angina, congestive heart failure exacerbation (New York Heart Association Classification ≥ Class II), or unstable cardiac arrhythmia (< 3 months prior to enrollment). Stable cardiac arrhythmia (such as atrial fibrillation, atrial flutter) controlled on or off medications is permitted.
16. Known additional malignancy that is progressing or has required active treatment within the past 2 years. Patients with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, low grade prostate cancer, carcinoma in situ (e.g., breast carcinoma in situ, bladder carcinoma in situ) that have undergone potentially curative therapy or are on active surveillance are not excluded. Patients with cancer not detectable on imaging, not receiving active treatment, and not expected to impact 5-year life expectancy are eligible to enroll.
17. Unable to swallow orally administered medication intact or has a history or current evidence of a gastrointestinal disorder (e.g., inflammatory bowel disease, Crohn's disease, ulcerative colitis, gastrectomy, partial bowel obstruction, malabsorption) or impaired liver function or diseases that in the opinion of the investigator may significantly alter the absorption and metabolism of oral medications.
18. History or evidence of any other clinically unstable/uncontrolled disorder, condition, or disease (including, but not limited to, cardiopulmonary, renal, metabolic, hematologic, or psychiatric) other than their primary malignancy, that in the opinion of the investigator would pose a risk to patient safety or interfere with study evaluations, procedures, or completion.
19. Known allergy or hypersensitivity to any component or formulation components of retifanlimab and ruxolitinib.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-08 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Recommended phase 2 dose | 28 days
  Determine the recommended phase 2 dose of ruxolitinib in combination with a fixed dose of retifanlimab. The recommended phase 2 dose will be determined by assessment of the dose limiting toxicities during the first cycle of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Rana McKay, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego Moores Cancer Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No